CLINICAL TRIAL: NCT02074579
Title: A Phase 2, Single-center, Randomized, Double-Blinded, Placebo-Controlled Study on the Efficacy of Daikenchuto (TU 100) to Relieve Abdominal Bloating in Female Subjects With Irritable Bowel Syndrome
Brief Title: A Safety and Efficacy Study of Daikenchuto (TU-100) to Relieve Abdominal Bloating in Female Subjects With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tsumura USA (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TU100CPT6
Record Dates: First submitted 2014-02-24; First posted 2014-02-28 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Irritable Bowel Syndrome in Females
Keywords: Irritable Bowel Syndrome; Rome III criteria; abdominal bloating; natural; herbal; Kampo; Adult ages 18 to 65; Female subjects
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine; dai-kenchu-to

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TU-100 (Experimental): 15g TU-100 (oral, daily) for 4 consecutive weeks (administered as 5g three times daily)
  Interventions: Drug: TU-100
- Matching placebo (Placebo Comparator): Matching placebo given 5g three times daily orally for 4 consecutive weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TU-100 — 15g daily, orally as 5g three times daily for 4 consecutive weeks
  Other Names: Daikenchuto
  Arms: TU-100
Drug: Placebo — Matching placebo given 5g three times daily orally for 4 consecutive weeks
  Arms: Matching placebo

SUMMARY:
The aim of this study is to assess the effect of orally administered TU-100 (5 g three times daily [TID]) as compared to placebo on abdominal bloating rating in female IBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet Rome III criteria for IBS (any subtype)
* Female aged 18 to 65 years, inclusive
* If of childbearing potential, prepared to use suitable forms of contraception throughout the study and for 30 days after the last dose i.e., hormonal contraceptives (such as oral contraceptives, Depo-Provera, NuvaRing, Essure), condoms used with a spermicide, an intrauterine device, or abstinence. Females are not considered to be of childbearing potential if they are naturally postmenopausal (no menses for at least 1 year and, if < 55 years of age, have a documented follicle-stimulating hormone [FSH] level of ≥ 35 mIU/mL) or have documentation of surgical sterility
* Have a BMI between 18 and 30 kg/m2, inclusive
* Have a negative pregnancy urine screening at Visit 1, if of childbearing potential
* Able to provide written consent
* Able to take oral administration of the testing medications
* Have a self-reported average abdominal bloating rating (>3 daily ratings over the preceding 7 days) equal or greater than 4 on a numerical scale of 0 to 20.

Exclusion Criteria:

* Have a structural or metabolic disease or condition that affects the GI system, excluding asymptomatic gallstones or uncomplicated gastroesophageal reflux disease, or any medical condition that may be a cause of constipation or diarrhea (e.g., hypothyroid status, poorly controlled diabetes, diabetic neuropathy or autonomic neuropathy)
* Be taking any medication that, in the opinion of the Principle Investigator (PI), has potential to alter GI transit. A full list of prohibited medications is provided in the protocol. Have history or presence of any chronic lung disease
* Have presence of hepatic dysfunction, jaundice, or abnormal serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values exceeding 2.5 x upper limit of normal
* Currently pregnant or lactating
* Have a positive urine drug test at screening (subjects who initially test positive will be allowed one retest)
* Be a known substance abuser or be considered to be an alcoholic not in remission
* Have participated in another clinical study in the past 30 days
* Use of supplemental ginger, ginseng, or Zanthoxylum fruit for 2 weeks prior to randomization and throughout the course of the study.
* Have a history of allergic reaction to ginseng, ginger or Zanthoxylum fruit
* Be clinically lactose-intolerant
* Have any other condition that, in the opinion of the PI, causes the subject to be unsuitable to participate
* Have taken antibiotics in the last 3 months
* Have had gastroenteritis ("stomach flu") in the last 3 months
* Have taken probiotics in the last 3 months (over-the-counter [OTC] products or supplements only; food products such as yogurts are permitted).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Abdominal bloating rating | 4 weeks
  Change in abdominal bloating rating, through comparison of the change in average ratings from the 7 days prior to baseline (Visit 2) to the last 7 days of the 4 week treatment period (Visit 4), between TU-100 15 g and placebo.

SECONDARY OUTCOMES:
AUC for abdominal bloating ratings using lactulose challenge | Baseline and 4 weeks
  Change in area under the curve (AUC) for abdominal bloating ratings obtained during the lactulose challenge at Visit 2 (baseline) and at Visit 4 (4 weeks). The data are collected at -0.5, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8 hours after taking test meal (lactulose).
Abdominal bloating ratings | 4 weeks
  Change in the average of abdominal bloating ratings from the 7 days prior to baseline to the 7 days prior to Visit 3 (2 weeks) and to Visit 5 (8 weeks)
Overall IBS Severity | 4 weeks
  Change in Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) total score from baseline to Visits 3, 4, and 5
GI symptom ratings | 4 week
  Change in the average of GI symptom ratings from the 7 days prior to baseline to the 7 days prior to Visit 3 and to Visit 5
Quality of Life effect | 4 weeks
  Change in IBS-QOL score from baseline to Visits 3, 4, and 5
Mood symptom ratings | 4 weeks
  Change in the average of mood symptom ratings from the 7 days prior to baseline to the 7 days prior to Visit 3 and to Visit 5

OTHER OUTCOMES:
Physical Examination | 4 weeks
  Physical examination at Visits 1, 2 and 4
Vital Signs | 4 weeks
  2. Vital signs (pulse, blood pressure, temperature, and respiration rate) at Visits 1, 2 and 4
Adverse Events and Concomitant Medications | 8 weeks
  Interview for adverse events (AEs) and concomitant medications at Visits 3, 4 and 5
Laboratory safety tests | 8 weeks
  Laboratory safety tests including hematology, chemistry, and urinalysis at Visits 1, 2 and 4. Pregnancy test for subjects of childbearing potential at Visits 1, 2, 3, 4 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tillisch, MD, Principal Investigator — Oppenheimer Family Center of Neurobiology of Stress, UCLA
Locations (1):
- Oppenheimer Family Center for Neurobiology of Stress Division of Digestive Diseases David Geffen School of Medicine at UCLA, Los Angeles, California, United States